CLINICAL TRIAL: NCT00282503
Title: A Randomized, Controlled, Parallel-Group, Multicenter Study of Extracorporeal Photoimmune Therapy With THERAKOS* UVADEX* for the Treatment of Patients With Newly Diagnosed Acute Graft Versus-Host Disease
Brief Title: Extracorporeal Photoimmune Therapy With UVADEX for the Treatment of Acute Graft Versus-Host Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Mallinckrodt (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Acute GvHD-1
Record Dates: First submitted 2006-01-24; First posted 2006-01-26 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Acute Graft-versus-Host Disease
Keywords: aGvHD
MeSH Terms: interventions — Methylprednisolone; Eosinophil Cationic Protein

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- methylprednisolone equivalent. (Active Comparator): 2mg/kg daily will be administered initially and may be tapered according to a tapering schedule provided in the protocol.
  Interventions: Drug: Methoxsalen+ECP, Methylprednisolone
- Uvadex+ECP (Experimental): Those patients randomized to the ECP Treatment arm will receive ECP treatments by the following regimen:
  * Weeks 1 through Week 3 - 3 times within each week. (Treatments do not have to be performed on consecutive days but should be completed within the 7-day period),
  * Weeks 4 through 12 - 2 times each week. (It is preferable that patients receive ECP treatments on consecutive days
  Interventions: Drug: Methoxsalen+ECP, Methylprednisolone; Procedure: Ecp

INTERVENTIONS:
Drug: Methoxsalen+ECP, Methylprednisolone — Those patients randomized to the ECP Treatment arm will receive ECP treatments by the following regimen:
  * Weeks 1 through Week 3 - 3 times within each week. (Treatments do not have to be performed on consecutive days but should be completed within the 7-day period),
  * Weeks 4 through 12 - 2 times each week. (It is preferable that patients receive ECP treatments on consecutive days within a week, but there should never be > 4 days between the ECP treatments within a week.)
  Methylprednisolone will be started at 2mg/kg daily dose and may be tapered by reducing dose each week at the following reductions:
  Daily Dose (mg/kg)
  1 1.5 2 1.0 3 0.70 4 0.50 5 0.40 6 0.30 7 0.20 8 0.10
  Other Names: Uvadex+ ECP
Procedure: Ecp — ECP or Extra Corporeal Phototherapy will be used with UVADex
  Arms: Uvadex+ECP

SUMMARY:
The purpose of this study is to compare the safety and efficacy of ECP treatment combined with high dose corticosteroids versus high dose corticosteroids alone, in the treatment of patients with newly diagnosed acute GvHD (Grades II to III) that developed within 100 days following an allo HPCT.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to conducting any study procedure.
2. Patients must be greater than or equal to 18 years old and weigh greater than or equal to 40 kg (88 lb).
3. Patients must have received an allogeneic hematopoietic BMT or PBSCT with myeloablative or reduced-intensity conditioning and have a new onset of acute GvHD, Grades II to III, which includes the skin and developed within 100 days following an allo-HPCT.
4. Patients must have received an allogeneic hematopoietic BMT or PBSCT from a related or unrelated donor that is matched at a minimum at the HLA-A, -B, and -DR loci (i.e., at least a 6 out of 6 match). HLA-A and -B match should be determined by serologic testing, and HLA-DR should be matched by molecular methods.
5. Patients must be receiving only a calcineurin inhibitor at study entry as part of their acute GvHD prophylactic regimen. Patients may have received additional immunosuppressants for acute GvHD prophylaxis prior to study entry.
6. Patients must have a Karnofsky performance greater than or equal to 50.
7. Patients must be able and willing to comply with all study procedures.
8. Patients must receive, or must have received, the first corticosteroid dose of approximately 2.0 mg/kg/day but no more than 2.5 mg/kg/day (methylprednisolone equivalent) within 24 hours of the initial diagnosis of Grade II to III acute GvHD. (Up to 2.5 mg/kg/day is allowed for inadvertent dosing fluctuations for reasons other than lack of response.)
9. Female patients must be one of the following: postmenopausal, surgically incapable of bearing children, practicing an acceptable method of birth control (acceptable methods include hormonal contraceptives, intrauterine device, and spermicide and barrier). Abstinence or partner/spouse sterility may also qualify at the Investigator's discretion. If a female patient is of childbearing potential, she must have a negative urine pregnancy test at screening. Male patients must also commit to using adequate contraceptive precautions (condoms). All patients (both males and females of childbearing potential) must commit to using adequate contraceptive precautions throughout their participation in the study and for at least 3 months following their last ECP treatment.

Exclusion Criteria:

1. Patients who have been diagnosed with chronic GvHD, including de novo chronic GvHD, prior to 100 days following an allo-HPCT.
2. Patients who have received donor lymphocyte infusions.
3. Patients with uncontrolled life-threatening infections.
4. Patients who have a white blood cell (WBC) count < 1.5 x 10^9/L (1,500/mcL).
5. Patients who have a platelet count < 20.0 x 10^9/L (20,000/mcL), despite platelet transfusion.
6. Patients whose total bilirubin is greater than or equal to 22 mg/dL.
7. Patients who have an International Normalized Ratio (INR) greater than or equal to 2.
8. Patients who are enrolled in any concomitant investigation for the treatment of acute GvHD.
9. Patients who are unable to tolerate the extracorporeal volume shifts associated with ECP treatment due to the presence of any of the following conditions: uncompensated congestive heart failure, pulmonary edema, severe chronic obstructive pulmonary disease, severe asthma, renal failure, hepatic encephalopathy, or hepatorenal syndrome.
10. Female patients whose hemoglobin (Hgb) is < 8.5 g/dL or male patients whose Hgb is < 10.0 g/dL at screening, despite packed red blood cell transfusion.
11. Patients who have a poor tolerability of venipuncture or a lack of adequate venous access for required treatments and blood sampling.
12. Patients who have a known hypersensitivity or allergy to Oxsoralen (methoxsalen).
13. Patients who have a known hypersensitivity or allergy to both heparin and citrate products.
14. Female patients who are pregnant and/or lactating.
15. Patients who have co-existing melanoma, basal cell or squamous cell skin carcinoma, aphakia, photosensitive disease (e.g., porphyria, systemic lupus erythematosus, or albinism), white blood cell count > 25,000 cells/mm3, previous splenectomy, or coagulation disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To compare the safety and efficacy of ECP treatment combined with high dose corticosteroids versus high dose corticosteroids alone, in patients with newly diagnosed acute GvHD (Grades II to III) that developed within 100 days following an allo HPCT. | 8 weeks
  The primary efficacy analysis will be performed on the primary endpoint. The primary efficacy variable in this study is complete resolution of acute GvHD, defined as less than Grade I acute GvHD, according to the Glucksberg-Seattle criteria.

CONTACTS AND LOCATIONS:
Locations (35):
- United States (5):
  - University of Florida, Gainesville, Florida
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Weill Medical College of Cornell University, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Leukemia and Bone Marrow Transplant Center - Avera Cancer Institute, Sioux Falls, South Dakota
- Australia (3):
  - Royal Brisbane Women's Hospital, Brisbane
  - Saint Vincent's Hospital, Darlinghurst
  - Westmead Hospital, Westmead
- Medical University of Vienna, Vienna, Austria
- Belgium (3):
  - Universite Catholique De Louvain, Brussels
  - University Hospital Gasthuisberg, Leuven
  - Centre Hopitalier Universitaire Sart Tilman Liege, Liège
- Canada (4):
  - Vancouver General Hopsital, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hopital, Montreal
  - Royal Victoria Hospital, Montreal
- France (2):
  - Centre Hospitalier Universitaire Hospital Bordeaux, Bordeaux
  - St. Louis Hospital, Paris
- Germany (10):
  - University of Koln, Cologne
  - University of Dresden, Dresden
  - Klinikum der Universitat Erlangen-Nurnberg, Erlangen
  - Universitats Hautklinik, Essen
  - Universitatskrankenhaus Hamburg-Eppendorf, Hamburg
  - Universitatsklinikum Leipzig, Leipzig
  - Ludwig-Maximillians-Universitat Munchen, München
  - Universitat Regensburg, Regensburg
  - University of Rostock, Rostock
  - Stammzelltransplantationzentrum der Universitat Wurzbrug, Würzburg
- Italy (2):
  - Universita di Siena Policlinico Le Scotte, Siena, Sienna
  - San Martino Hospital, Genova
- Utrecht University Medical Center, Utrecht, Netherlands
- Kantonsspital Basel, Basel, Switzerland
- United Kingdom (3):
  - Hammersmith Hospital, London
  - Royal Victoria Infirmary, Newcastle
  - Rotheram General Hospital, Rotheram Yorkshire